CLINICAL TRIAL: NCT05216744
Title: Comparison of Efficacy of Two Combination Regimens for the Treatment of Uncomplicated Neisseria Gonorrhoeae and Chlamydia Trachomatis Coinfection
Brief Title: Comparison of Efficacy of Two Combination Regimens for the Neisseria Gonorrhoeae and Chlamydia Coinfection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haiphong University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPMU.19.10.21
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-01

CONDITIONS: Neisseria Gonorrhoeae Infection; Chlamydia Trachomatis Infection
Keywords: Neisseria Gonorrhoeae; Chlamydia Trachomatis; reinfection
MeSH Terms: conditions — Gonorrhea; Reinfection | interventions — Ceftriaxone; Doxycycline; Cefixime

STUDY DESIGN:
Intervention Model Description: Each subject will receive one of two combination regimens including regimen A (Doxycycline plus Cefixime) or regimen B (Doxycycline plus Ceftriaxone).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycycline plus ceftriaxone (Experimental): Each subject will receive 100 mg doxycycline twice daily for seven days and a single dose of ceftriaxone 1000 mg intravenously
  Interventions: Drug: Ceftriaxone 1000mg + doxycycline 100 mg
- Doxycycline plus cefixime (Active Comparator): Each subject will receive 100 mg doxycycline twice daily for seven days and a single oral dose of cefixime 800 mg
  Interventions: Drug: Cefixime 800mg + doxycycline 100 mg

INTERVENTIONS:
Drug: Ceftriaxone 1000mg + doxycycline 100 mg — Study comparing the effectiveness of two combination regimens in the treatment of gonorrhea and chlamydia, including regimen A (100mg doxycycline orally twice a day for 7 days + 1 dose of 1000mg ceftriaxone intravenously) and regimen B (100mg doxycycline). orally for 7 days + 1 oral dose of 800mg cefixime)
  Other Names: Ceftriaxone 1000mg IV plus doxycycline 100 mg PO twice daily in 7 days
  Arms: Doxycycline plus ceftriaxone
Drug: Cefixime 800mg + doxycycline 100 mg — Study comparing the effectiveness of two combination regimens in the treatment of gonorrhea and chlamydia, including regimen A (100mg doxycycline orally twice a day for 7 days + 1 dose of 1000mg ceftriaxone intravenously) and regimen B (100mg doxycycline). orally for 7 days + 1 oral dose of 800mg cefixime)
  Other Names: a single oral dose of Cefixime 800mg plus doxycycline 100 mg PO twice daily in 7 days
  Arms: Doxycycline plus cefixime

SUMMARY:
The frequency of Chlamydia trachomatis and Neisseria gonorrhoeae coinfection can vary depending on their individual incidence and prevalence rates.Single-agent therapy with ceftriaxone is the preferred regimen for treatment of gonococcal infections. If an injectable cephalosporin is not available, cefixime is the only oral cephalosporin that can be used for gonococcal therapy. Doxycycline was recommended for presumptive treatment of chlamydia in nonpregnant individuals with gonococcal infection. The study is conducted to evaluate the effectiveness of two regimens in combination with doxycycline with cefixime or ceftriaxone.

DETAILED DESCRIPTION:
Gonococcal infections, including urethritis, cervicitis, epididymitis, and proctitis, are a significant cause of morbidity among sexually active men and women. The treatment of these sexually transmitted infections (STIs) has evolved over the years, mainly due to the emergence of antibiotic resistance. The frequency of Chlamydia trachomatis and Neisseria gonorrhoeae coinfection can vary depending on their individual incidence and prevalence rates. Ceftriaxone is highly effective against susceptible N. gonorrhoeae. Single-agent therapy with ceftriaxone is the preferred regimen for treatment of gonococcal infections. These doses of ceftriaxone are higher than previously recommended due to concerns regarding rising gonococcal minimum inhibitory concentrations (MICs) worldwide. If an injectable cephalosporin is not available, cefixime is the only oral cephalosporin that can be used for gonococcal therapy. Doxycycline (100 mg orally twice daily for seven days) was recommended for presumptive treatment of chlamydia in nonpregnant individuals with gonococcal infection. The study is conducted to evaluate the effectiveness of two regimens in combination with doxycycline with cefixime or ceftriaxone.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 ages with laboratory-documented uncomplicated Chlamydia trachomatis and Neisseria gonorrhoeae reinfection at any site

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Hypersensitivity to cephalosporins or penicillins
* significant renal failure or hepatic failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
cure rate | 5th day after treatment
  a negative test of cure for Chlamydia trachomatis and Neisseria gonorrhoeae

SECONDARY OUTCOMES:
Side effects | From 1st day of study to 5th day after treatment
  Any side effects from interventions in two arms

CONTACTS AND LOCATIONS:
Overall Officials: Phuong Nguyen, PhD, Study Director — Hai Phong University of Medicine and Pharmacy
Locations (1):
- Haiphong International Hospital, Haiphong, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen PTT, Pham HV, Van DH, Pham LV, Nguyen HT, Nguyen HV. Randomized controlled trial of the relative efficacy of high-dose intravenous ceftriaxone and oral cefixime combined with doxycycline for the treatment of Chlamydia trachomatis and Neisseria gonorrhoeae co-infection. BMC Infect Dis. 2022 Jul 9;22(1):607. doi: 10.1186/s12879-022-07595-w. PMID 35810277